CLINICAL TRIAL: NCT03498378
Title: A Phase I Study of Avelumab, Palbociclib, and Cetuximab in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Avelumab, Cetuximab, and Palbociclib in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kathryn Gold (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Kathryn Gold, Assistant Clinical Professor of Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 171386
Record Dates: First submitted 2018-03-27; First posted 2018-04-13 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Avelumab; Palbociclib; Cetuximab; Head and Neck Squamous Cell Carcinoma; cancer; Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — avelumab; palbociclib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Avelumab, Palbociclib, and Cetuximab (Experimental): Identify the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) for the combination of palbociclib, avelumab, and cetuximab
  Interventions: Drug: Avelumab; Drug: Palbociclib; Drug: Cetuximab

INTERVENTIONS:
Drug: Avelumab — Avelumab (IV on days 1 and 15 of 28 day cycle)
  Other Names: Bavencio
Drug: Palbociclib — Palbociclib (PO daily, days 1-21 of 28 day cycle)
  Palbociclib will be administered in capsules of 125 mg, 100 mg, and 75 mg, depending on dosage. Patients will be instructed to take their assigned dose once daily with food for 21 days followed by 7 days off therapy. Patients will be encouraged to take their dose at approximately the same time each day.
  Other Names: IBRANCE
Drug: Cetuximab — Cetuximab (IV 400 mg/m2 x 1, then weekly)
  Cetuximab is administered intravenously once weekly via infusion pump or syringe pump with infusion rate not to exceed 10 mg/min.
  Other Names: ERBITUX

SUMMARY:
The purpose of the study is to find out if the study drugs Avelumab, Cetuximab, and Palbociclib will slow or stop your cancer from getting worse, and whether it causes side effects. The second purpose is to measure whether your cancer responds to the study drugs Avelumab, Cetuximab, and Palbociclib. The study drugs Avelumab, Cetuximab, and Palbociclib are types of drugs called a monoclonal antibody. Monoclonal antibodies are made to recognize, target, and bind to specific proteins on cells the building blocks making up your tissues.

DETAILED DESCRIPTION:
This is an open-label phase I trial with a 3+3 dose escalation design. All patients will receive avelumab, cetuximab, and palbociclib. This study will enroll patients with head and neck squamous cell carcinoma not amenable to curative intent therapy.

Treatment will be administered in 28 day cycles with a pre-defined dose escalation schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of the head and neck not amenable to curative intent therapy.
* Presence of measurable tumor lesions per RECIST criteria v1.1
* Life expectancy greater than 12 weeks.
* Adequate hematologic, hepatic, and renal function
* Negative serum or urine pregnancy test for women of child bearing potential

Exclusion Criteria:

* Prior therapy with an EGFR inhibitor or PD-1 or PD-L1 inhibitor in the recurrent or metastatic setting
* Uncontrolled central nervous system metastases (stable metastases permitted)
* Chemotherapy 28 days prior to first administration of study treatment and/or monoclonal antibody ≤8 weeks prior to first administration of study treatment.
* History of other malignancies,
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration of >10 mg/day of prednisone or equivalent)
* Prior organ transplantation
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 12 months
  maximum tolerated dose/recommended phase II dose.

SECONDARY OUTCOMES:
Overall response rate | through study completion, an average of 3 years
  Determined by RECIST 1.1
progression free survival | through study completion, an average of 3 years
  progression free survival
overall survival | through study completion, an average of 3 years
  overall survival
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Gold, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dennis MJ, Sacco AG, Qi Y, Bykowski J, Pittman E, Chen R, Messer K, Cohen EEW, Gold KA. A phase I study of avelumab, palbociclib, and cetuximab in patients with recurrent or metastatic head and neck squamous cell carcinoma. Oral Oncol. 2022 Dec;135:106219. doi: 10.1016/j.oraloncology.2022.106219. Epub 2022 Oct 21. PMID 36279618